CLINICAL TRIAL: NCT06198608
Title: Interstitial Lung Disease Misdiagnosis in Cardiac Patients
Brief Title: Misdiagnosis Between Interstitial Lung Disease and Cardiac Patients
Status: Unknown | Type: Observational
Last Known Status: Not yet recruiting
Sponsor: Assiut University (Other)
Responsible Party: Principal Investigator, Hend Mohamed Sayed Mohamed, doctor, Assiut University
Other Study IDs: ILD&Cardiac patient
Record Dates: First submitted 2023-12-26; First posted 2024-01-10 (Actual); Last update posted 2024-01-10 (Actual); Status verified 2023-12

CONDITIONS: ILD

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
Aim of the study To determine the frequency misdiagnosis of cardiac congestion as interstitial lung disease based on initial High Resolution CT interpretation alone.

To identify specific HRCT findings that are more commonly associated with misdiagnosis versus correct diagnosis of the underlying condition.

To establish diagnostic criteria or HRCT patterns that distinguish cardiac congestion from interstitial lung disease

DETAILED DESCRIPTION:
Observational study of 150 patients found that cardiac congestion was misdiagnosed as interstitial lung disease in 24% of cases on initial HRCT imaging alone. Echocardiography and clinical correlation were needed to make the correct diagnosis .

Misdiagnosis can lead to inappropriate treatment with immunosuppressive drugs which could exacerbate right heart failure in patients who actually have cardiac congestion. Correct diagnosis is important for prognosis and management.

Subtle findings like upper lobe predominance of opacities, septal lines and a mosaic attenuation pattern on HRCT favor interstitial lung disease, while diffuse ground glass with central and perihilar distribution favors cardiac congestion .

Associated findings on HRCT like enlarged cardiac silhouette, pleural and pericardial effusions help suggest the diagnosis of cardiac congestion over idiopathic interstitial pneumonia .

Integrating clinical data on risk factors for heart failure, echocardiography findings and follow-up imaging response to diuretic therapy can help differentiate the two conditions when HRCT is non-specific

ELIGIBILITY:
Inclusion Criteria:

* Patients who underwent HRCT imaging of the chest for evaluation of suspected interstitial lung disease
* Initial radiology report included a definitive diagnosis of interstitial lung disease patterns
* Age 18+ years
* No prior history of pulmonary or cardiac

Exclusion Criteria:

* Inconclusive or unclear initial HRCT report
* Underlying diagnosis other than interstitial lung disease or cardiac congestion

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: prospective observational study design. Inclusion of patients who underwent HRCT for suspected interstitial lung disease or cardiac congestion.
  HRCT scans by experienced radiologists who are blinded to the initial interpretation and final diagnosis.
  Development of specific diagnostic criteria or guidelines to differentiate between interstitial lung disease and cardiac congestion based on HRCT findings.
  Collection of echocardiogram,lab results, clinical follow up to determine finial diagnosis.
  Comparison of Initial HRCT Interpretation: Comparison of the initial HRCT interpretation with the final diagnosis to determine the rate of misdiagnosis.
Sampling Method: Probability Sample
Enrollment: 80 (Estimated)
Dates: Start 2024-01-01 (Estimated); Primary Completion 2024-11-01 (Estimated); Study Completion 2024-12-30 (Estimated)

PRIMARY OUTCOMES:
Accuracy of initial HRCT interpretation | baseline
  (percentage of cases initially read as interstitial lung disease that were later found to be cardiac congestion)

SECONDARY OUTCOMES:
Time to correct diagnosis | baseline
  Mean or median number of days/months between initial misdiagnosis on HRCT and reaching accurate diagnosis of cardiac congestion

CONTACTS AND LOCATIONS:
Overall Officials: marwan sayed, MD, Study Chair — lecture in cardiac diseases; samaa elkossi, MD, Study Chair — Lecture inradiology departement

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Nathan SD, Pastre J, Ksovreli I, Barnett S, King C, Aryal S, Ahmad K, Fukuda C, Ramalingam V, Chung JH. HRCT evaluation of patients with interstitial lung disease: comparison of the 2018 and 2011 diagnostic guidelines. Ther Adv Respir Dis. 2020 Jan-Dec;14:1753466620968496. doi: 10.1177/1753466620968496. PMID 33121391
- [Background] Case AH, Beegle S, Hotchkin DL, Kaelin T, Kim HJ, Podolanczuk AJ, Ramaswamy M, Remolina C, Salvatore MM, Tu C, de Andrade JA. Defining the pathway to timely diagnosis and treatment of interstitial lung disease: a US Delphi survey. BMJ Open Respir Res. 2023 Nov 24;10(1):e001594. doi: 10.1136/bmjresp-2022-001594. PMID 38007235